CLINICAL TRIAL: NCT02388685
Title: Comprehensive Magnetic Resonance in Peripheral Arterial Disease.3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate patient recruitment
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher Kramer, Professor of Radiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-HSR# 16084
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; exercise; perfusion; energetics; magnetic resonance imaging; magnetic resonance spectroscopy
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home exercise (Experimental): Patients will undergo home exercise therapy under the supervision of the exercise laboratory
  Interventions: Other: Exercise
- No exercise (No Intervention): Patients will continue with usual care

INTERVENTIONS:
Other: Exercise — Home exercise therapy
  Arms: Home exercise

SUMMARY:
The goal is to test the ability to detect improved calf muscle perfusion and energetics in PAD patients in a randomized controlled trial of home exercise therapy. Eighty patients will be randomized to a 12 week home exercise program or no program (control).

DETAILED DESCRIPTION:
The goal is to test the ability to detect improved calf muscle perfusion and energetics in PAD patients in a randomized controlled trial of home exercise therapy. Eighty patients will be randomized to a 12 week home exercise program or no program (control). Patients will be studied before and after program completion with MRI/MRS, calf muscle biopsy for capillary density, and exercise performance measures. Arterial spin labeling peak exercise calf muscle perfusion will be used as the primary endpoint in the most symptomatic leg. All will undergo ASL, peak exercise PCr recovery kinetics, calf muscle biopsy, and functional measures including treadmill exercise, VO2 testing, and 6-minute walk. Correlations will be examined between changes in perfusion and energetics with changes in capillary density, peak VO2, and functional capacity from before to after completion of home exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented ABI 0.5-0.9
* Ability to walk on treadmill

Exclusion Criteria:

* Lower extremity vascular surgery, angioplasty or lumbar sympathectomy within 3 months of enrollment
* Critical limb ischemia
* Known or suspected peripheral neuropathy, heel cord contracture and foot deformity
* Other conditions that limit walking, e.g. lung disease or arthritis
* Active coronary artery disease such as unstable angina, significant left main disease or three vessel coronary artery disease (>70% stenosis, unprotected by grafts) or recent (<2 months) myocardial infarction,
* BMI > 40,
* Known contraindication to MRI (intracardiac pacer, defibrillator, certain intracranial aneurysm clips, intraocular or cochlear implants, claustrophobia, etc.)
* Allergy to lidocaine or xylocaine (local anesthetic)

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Exercise calf muscle perfusion | Change from baseline at 12 weeks
  Arterial spin labeling MRI at peak exercise
Exercise calf muscle energetics | Change from baseline at 12 weeks
  Phosphocreatine recovery kinetics by MR spectroscopy at end exercise

SECONDARY OUTCOMES:
Calf muscle capillary density | Change from baseline at 12 weeks
  Biopsy sample of calf muscle for capillary density
Treadmill testing | Change from baseline at 12 weeks
  Treadmill testing with peak VO2 measures
6-minute walk test | Change from baseline at 12 weeks
  6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Kramer, MD, Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States